CLINICAL TRIAL: NCT05239091
Title: Comparison of the Efficacy of Prolotherapy Injection Therapy and Local Anesthetic (Lidocaine) Injection Therapy in Myofascial Pain Syndrome.
Brief Title: Comparison of the Efficacy of Prolotherapy Injection Therapy & Local Anesthetic Injection Therapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Necat Akgun, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FTRinjection
Record Dates: First submitted 2022-01-24; First posted 2022-02-14 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2022-08

CONDITIONS: Myofascial Pain Syndrome of Neck
Keywords: Lidocaine; dextrose prolotherapy; pain
MeSH Terms: conditions — Pain | interventions — Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, triple blinded, clinical trials
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, Outcomes Assessor, and Investigator (statistician) will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextrose prolotherapy (Experimental): :%15 dextrose prolotherapy injection will be applied to trigger point
  Interventions: Drug: Dextrose solution
- Lidocaine (Active Comparator): %2 lidocaine injection will be applied to trigger point
  Interventions: Drug: Lidocain

INTERVENTIONS:
Drug: Dextrose solution — A total of 3 doses of dextrose prolotherapy will be administered with an interval of 2 weeks.
  Other Names: Dextrose prolotherapy
  Arms: Dextrose prolotherapy
Drug: Lidocain — A total of 3 doses of lidocaine will be administered with an interval of 2 weeks.
  Other Names: Local anesthetic
  Arms: Lidocaine

SUMMARY:
Myofascial pain syndrome is a disease characterized by pain over the trigger point in a taut muscle band. After the correct diagnosis is made, many treatment methods can be applied.

One of these treatments is the treatment with prolotherapy injection. Proliferant reveals defense mechanisms remove them and then start the healing process in the damaged area. Usually, dextrose water is used. Lidocaine is an anesthetic. With lidocaine injection, the passage of painful stimuli is prevented and the opioid system is activated. The aim of the study is to compare the efficacy of prolotherapy and lidocaine treatment in the myofascial pain syndrome.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study. The population of the study consists of volunteer patients who can apply to Istanbul Physical Therapy and Rehabilitation Training and Research Hospital, and meet the inclusion criteria. Twenty-eight people will be selected from the participants who volunteered for the study and will be divided into the study group and control groups with the permutation block randomization method. At the beginning, all patients will be asked about their gender, age, body mass index, education level, occupation, duration of complaint, previous treatments, and the last time received treatment.

Patients will be recruited equally to the control and study groups, with 14 patients in each group. 15% dextrose injection treatment will be applied to the study group. 2% lidocaine injection treatment will be applied to the control group. The subjects will be asked to sit on a chair and the trigger point will be determined in the upper trapezius muscle in both groups. A total of 3 sessions of injection treatment will be applied to the trigger points (at the beginning, at the 2nd, and 4th weeks). It will be planned to be 2 weeks between each injection session. 1 month after the third session injection, patients will be called for control purposes.

The application will be made using a 25 gauge injector. Before the injection, the skin will be cleaned with alcohol and then dried. All patients will be injected into the trigger points in the upper trapezius muscle. Trigger point injection, on the other hand, is the compression of the isolated skin with the help of the thumb and middle finger and advancing the needle into the muscle at a 90-degree angle. Before the injection, a puncture will be made to make sure the needle is not in the blood vessel. Some of the mixtures will be injected into the trigger point and the rest around the trigger point. The same injection technique will be applied in both the control and study groups. Measurements will be made at the beginning (week 0), week 2, and week 4 before and after the injection when they come to the 1-month control. Adverse events related to injections will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Primary myofascial pain syndrome (MAS) in the upper trapezius muscle
* At least one active myofascial trigger point in the upper trapezius muscle
* Patients with symptoms between 1 day and 2 months
* Age:18 to 65 years old
* Cases who did not receive any physical therapy or medication to relieve pain

Exclusion Criteria:

* Having a sensory defect in the area to be injected
* Active inflammatory, rheumatic, or infectious disease
* Peripheral nerve lesions such as polyneuropathy, radiculopathy
* Those who use anticoagulants, those with bleeding diathesis
* Patients whose skin surface is not intact in the area to be injected
* Patients diagnosed with fibromyalgia or other common musculoskeletal pain syndromes
* Patients with a history of panic attacks
* Those who are allergic to local anesthetic drug
* People showing symptoms of Covid-19
* Those who have had a trigger point injection in the last 6 months
* Those who are pregnant
* Those who have undergone vertebral or shoulder surgery in the last 1 year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | Change from baseline pressure pain threshold at 2,4,6 and 8 weeks.
  It will be measured by algometer. Its unit is kg/cm2

SECONDARY OUTCOMES:
Pain intensity | Change from baseline pain intensity score at 2,4,6 and 8 weeks.
  Pain intensity will be evaluated by using a visual analog scale (VAS).The maximum score is 10 points. A higher score indicates a worse pain level
Pain tolerance measurement | change from baseline pain tolerance at 2,4,6 and 8 weeks.
  A pressure of 2.5 kg/cm2 will be applied to the trigger point using an algometer (WAGNER -FPK20) and patients will be asked to express their pain intensity according to the visual analog scale (VAS) scale. All patients will be informed that VAS is 0 (no pain) and 10 (worst pain imaginable), and will be asked to indicate the point between 0 and 10 that can represent the severity of their pain.
SF-36 (Short Form-36) Survey | Change from baseline SF-36 Short Form Survey score at 8 week.
  The scale consists of 36 items and these provide the measurement of 8 dimensions. Instead of giving only a single total score, the scale gives a total score for each subscale separately. Subscales evaluate health on a scale of 0 to 100, with 0 indicating poor health and 100 indicating good health.

CONTACTS AND LOCATIONS:
Overall Officials: Fatmanur Kesiktaş, Prof, Study Director — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Hospital, Istanbul, Turkey (Türkiye)